CLINICAL TRIAL: NCT06463509
Title: Establishment and Standardization of a Platform for In-depth Tumour Profiling (TUPRO) in Patients With Advanced Melanoma - a Prospective, Multicentric HFV Research Project/Category A
Brief Title: Establishment and Standardization of a Platform for In-depth Tumour Profiling (TUPRO) in Patients With Melanoma
Acronym: TUPRO
Status: Completed | Type: Observational
Sponsor: Reinhard Dummer (Other)
Responsible Party: Sponsor-Investigator, Reinhard Dummer, Professor, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: TUPRO-Melanoma
Record Dates: First submitted 2024-05-15; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Establishment of an in-deepth tumor profiling platform — In-depth tumor profiling beyond genomics

SUMMARY:
TUPRO-Melanoma is the first project of the Tumour Profiler (TUPRO) research collaboration, which in the long-term aims to generate data that will help to understand and report the individual tumour biology and the clinical parameters for patients with advanced malignancies using innovative molecular technologies and computational analyses for in-depth molecular profiling. TUPRO-Melanoma is an exploratory project that aims to establish a comprehensive platform for in-depth tumour profiling in patients suffering from advanced melanoma. Aims of this platform are to establish logistics and algorithms for integrative analyses and discover new molecular biomarker profiles/patterns.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance status ≤2 (not bedridden for more than 50% of waking hours)
* Stage III or IV cutaneous melanoma, or rare melanoma subtypes at any stage that require systemic therapy
* Written informed consent according to national legal and regulatory requirements prior to any project specific procedures

Exclusion Criteria:

* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the sponsor-project leader or site project leader may interfere with the project or affect patient compliance
* Legal incompetence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced melanoma (stage III or IV cutaneous melanoma, or rare melanoma subtypes at any stage that require systemic therapy)
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Sample Processing and Report Generation | through study completion, an average of 1 year
  * Number of samples (with sufficient material and quality) made available for intended analysis per technology
  * Number of molecular summary reports (generated from the translational domain) that could be made available to the Tumour Board
  * Number (proportion) of cases in which the Tumour Board considers the molecular summary report as useful for making a treatment recommendation on a scale from zero (not useful at all) to five (very useful).
  * Number (proportion) of cases in which the treating physician considers the Tumour Board's recommendation as useful for making a treatment decision on a scale from zero (not useful at all) to five (very useful)
  * Types of molecular information and combinations of molecular information from the biotechnology domain that the pre-Tumour Board considers as useful for making a treatment recommendation beyond routine diagnostics (incl. routine pathology and NGS testing)
Classification of proposed treatment options (according to the one of the 7 categories below) | through study completion, an average of 1 year
  Select one of the following categories:
  * On-label treatment with molecular matched treatment (SwissMedic label as reference) +/- radiotherapy or chemotherapy;
  * Treatment with classical chemotherapy +/- radiotherapy (on label if label available);
  * Referral to a suitable clinical trial;
  * Off-label treatment (SwissMedic label as reference) with molecular matched treatment or immunotherapy +/- radiotherapy or chemotherapy;
  * Off-label treatment (authorization in countries with comparable control systems for medicinal products as defined by SwissMedic) with molecular matched treatment or immunotherapy +/- radiotherapy or chemotherapy;
  * Immunotherapy
  * No active anti-tumour treatment (best supportive care)
Classification of Tumour Board's recommendations according to ESCAT (categories below) | through study completion, an average of 1 year
  Select one of the categories below:
  * I-A: prospective, randomised clinical trials show the alteration-drug match in a specific tumour type results in a clinically meaningful improvement of a survival end point
  * II-A: retrospective studies show patients with the specific alteration in a specific tumour type experience clinically meaningful benefit with matched drug com pared with alteration-negative patients
  * III-A: clinical benefit demonstrated in patients with the specific alteration (as tiers I and II above) but in a different tumour type. Limited/absence of clinical evidence available for the patient-specific cancer type or broadly across cancer types
  * IV-A: evidence that the alteration or a functionally similar alteration influences drug sensitivity in preclinical in vitro or in vivo models
  * X: No evidence that the genomic alteration is therapeutically actionable
Time to first subsequent treatment (TTFST) | through study completion, at least 6 month of follow up
  - Time to first subsequent treatment (TTFST), incl. best supportive care
Time to first subsequent treatment (TTFST) ratio | through study completion, at least 6 month of follow up
  - Time to first subsequent treatment (TTFST) ratio (TTFST 2 / TTFST 1: TTFST 2 = TTFST on current project; TTFST 1 = TTFST on previous treatment [before entering the project])
Toxicity | through study completion, at least 6 month of follow up
  - Frequency (proportion) of patients terminating treatment due to toxicity
Survival | through study completion, at least 6 month of follow up
  - Overall survival (OS), calculated from registration until death due to any cause
Event free survival | through study completion, at least 6 month of follow up
  - Event free survival (EFS), defined as time to treatment failure or death
Radiological tumour response | through study completion, at least 6 month of follow up
  - Proportion of patients with a radiological tumour response (CR / PR) according to local standards and trial protocol (in case of referral or trial)

SECONDARY OUTCOMES:
Quality of life | through study completion, at least 6 month of follow up
  - Quality of Life using the Functional Assessment of Cancer Therapy - General - 7 Item Version (FACT-G7) questionnaire should be assessed during regular data collection (optional).
  Score range: 0-28. The higher the score, the better the Quality of life (QoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miglino N, Toussaint NC, Ring A, Bonilla X, Tusup M, Gosztonyi B, Mehra T, Gut G, Jacob F, Chevrier S, Lehmann KV, Casanova R, Jacobs A, Sivapatham S, Boos L, Rahimzadeh P, Schuerch M, Sobottka B, Chicherova N, Yu S, Wegmann R, Mena J, Milani ES, Goetze S, Esposito C, Sarabia Del Castillo J, Frei AL, Nowak M, Irmisch A, Kuipers J, Baciu-Dragan MA, Ferreira PF, Singer F, Bertolini A, Prummer M, Lischetti U; Tumor Profiler Consortium; Aebersold R, Bacac M, Maass G, Moch H, Weller M, Theocharides APA, Manz MG, Beerenwinkel N, Beisel C, Pelkmans L, Snijder B, Wollscheid B, Heinzelmann V, Bodenmiller B, Levesque MP, Koelzer VH, Ratsch G, Dummer R, Wicki A. Feasibility of multiomics tumor profiling for guiding treatment of melanoma. Nat Med. 2025 Jul;31(7):2430-2441. doi: 10.1038/s41591-025-03715-6. Epub 2025 May 27. PMID 40425842